CLINICAL TRIAL: NCT00574158
Title: Project 2: Genetic Regulation of Ozone Induced Inflammation in Humans.
Brief Title: Pathogenesis and Genetics of Environmental Asthma Ozone Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Michael Foster, Professor, National Institute of Environmental Health Sciences (NIEHS)
Other Study IDs: 12496-CP-004; ES012496
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Asthma; Inflammation
Keywords: ozone; inflammatory airway disease; polymorphisms
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, and ebc collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
The goals of the research are designed to accomplish genetic association studies of candidate genes in healthy normal individuals exposed to 0.2 ppm for 2.25 hours with intermittent exercise in order to search for associations between defined genotypes/haplotypes and 3 specific in vivo respiratory endpoints: a) change in FEV1 immediately after ozone exposure; b) change nonspecific bronchial reactivity as reflected in the change in methacholine PC20 FEV1 24 hours after ozone exposure ; and c) change in lung epithelial integrity as reflected in the Clearance Halftime of technetium 24 hours after ozone exposure. These studies have been carried forward to take place in 4 phases:

i) healthy individuals have been exposed to O3 using our standard exposure protocol; and we will increase the numbers of individuals available for study.

ii) perform genetic association studies for the endpoints of spirometry (FEV1, FVC, FEV1/FVC), PC20 FEV1 for methacholine, and epithelial integrity (Clearance Halftime) for 3 candidate O3 response genes taken from literature searches and/or previously characterized to demonstrate associations. These physiologic endpoints have been examined in terms of both a continuum of response, and discrete "responder" and "non-responder" endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal lung function values, and of normal body habitus (i.e., < BMI of 30);
* Do not have a history of lung disease, and not taking any medications for lung disease or other clinical disorders, and no prior or current smoking history.

Exclusion Criteria:

* Non-willingness to sign a consent form for participation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults, 18-35 y of age, both genders.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2005-07; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pathogenesis and genetics of environmental asthma ozone study | acute and at 18 to 24 hour followup.
  Phenotype physiologic responses to ambient level of ozone exposure.

CONTACTS AND LOCATIONS:
Overall Officials: W Michael Foster, PhD, Principal Investigator — Duke University
Locations (1):
- W Michael Foster, PhD, Durham, North Carolina, United States

REFERENCES:
- [Derived] Hussain S, Johnson CG, Sciurba J, Meng X, Stober VP, Liu C, Cyphert-Daly JM, Bulek K, Qian W, Solis A, Sakamachi Y, Trempus CS, Aloor JJ, Gowdy KM, Foster WM, Hollingsworth JW, Tighe RM, Li X, Fessler MB, Garantziotis S. TLR5 participates in the TLR4 receptor complex and promotes MyD88-dependent signaling in environmental lung injury. Elife. 2020 Jan 28;9:e50458. doi: 10.7554/eLife.50458. PMID 31989925